CLINICAL TRIAL: NCT01889459
Title: Patient Registry of Percutaneous Coronary Intervention (PCI) for Chronic Total Occlusion (CTO) by Japanese Experts
Brief Title: Japanese CTO PCI Expert Registry
Status: Recruiting | Type: Observational
Sponsor: Kurashiki Central Hospital (Other)
Collaborators: Japanese CTO PCI Expert Registry investigators (Unknown)
Responsible Party: Sponsor
Other Study IDs: J-CTOPCI-ER2013
Record Dates: First submitted 2013-06-26; First posted 2013-06-28 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-07

CONDITIONS: Chronic Total Occlusion of Coronary Artery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- PCI for CTO

SUMMARY:
The purpose of this study is to establish a consensus of treatment strategy of percutaneous coronary intervention (PCI) for chronic total occlusion (CTO) through patient registry of PCI for CTO performed by Japanese certified operators.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for PCI

Patients who underwent PCI for CTO lesions that contain the following:

1. Thrombolysis in myocardial infarction trial (TIMI) 0
2. The occlusive period more than 3 months or unknown
3. The main coronary arteries (segment 1-3, 5-8, 11, 13), branches that have large perfusion area (segment 4PL, 9/10, 12) and graft

Exclusion Criteria:

Patients ineligible for PCI judged in clinical practice

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent PCI for CTO lesions by Japanese certified operators
Sampling Method: Probability Sample
Enrollment: 19000 (Estimated)
Dates: Start 2013-07; Primary Completion 2022-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
successful revascularization without any major adverse cardiocerebral events (MACCE) at early follow-up and MACCE during the 5-year follow-up | within the first 1 month (plus 1 month) after PCI and during the 5-year follow-up
  early and late results on major adverse cardiocerebral events (MACCE): all-cause death, coronary artery bypass grafting, re-PCI (target lesion revascularization/target vessel revascularization), admission for heart failure, myocardial infarction, admission for unstable angina, cerebrovascular disease, stent thrombosis in 19000 patients in and outside Japan

CONTACTS AND LOCATIONS:
Locations (1):
- Kurashiki Central Hospital, Kurashiki, Japan